CLINICAL TRIAL: NCT00725829
Title: Effects of Simvastatin Versus Simvastatin Combined With Ezetimibe on Blood Coagulation in Patients With Acute Coronary Events: Relationship With Cholesterol-Lowering and Anti-Inflammatory Properties
Brief Title: Hypolipemic Treatment in Acute Coronary Syndrome (ACS): Antithrombotic Effects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jagiellonian University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Anetta Undas, Jagiellonian University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Prot. 116
Record Dates: First submitted 2008-07-07; First posted 2008-07-31 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Acute Coronary Syndrome
Keywords: coagulation; cholesterol; acute ischemia; fibrin clot
MeSH Terms: conditions — Acute Coronary Syndrome; Thrombosis | interventions — Simvastatin; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): simvastatin 40g + ezetimibe 10g once a day
  Interventions: Drug: simvastatin; Drug: ezetimibe
- 2 (Placebo Comparator): simvastatin 40g + placebo once a day
  Interventions: Drug: simvastatin; Drug: placebo

INTERVENTIONS:
Drug: simvastatin — Simvastatin 40mg/d
Drug: ezetimibe — ezetimibe 10mg/d
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
The aim of the current study is to evaluate whether treatment with high doses of simvastatin can reduce coagulation activation in patients with acute coronary syndromes and if ezetimibe in conjunction with simvastatin may affect blood clotting in a similar manner.

The investigators hypotheses are as follows:

1. Intensive lipid lowering treatment with simvastatin (40 mg/day) and simvastatin (40 mg/day) combined with ezetimibe (10 mg/day) initiated after acute coronary syndrome leads to attenuation of blood coagulation including reduced thrombin generation, thrombin-mediated coagulant reactions, and improved structure of plasma clots.
2. Anticoagulant effects of simvastatin are weaker than those observed during administration of simvastatin and ezetimibe.

DETAILED DESCRIPTION:
Clinical status will be evaluated during hospitalization, and then on the out-patient basis. All cardiovascular events (fatal or nonfatal myocardial infarction, unstable angina, sudden cardiac death, all-cause death, stroke, TIA) will be recorded and the patients who underwent acute PCI will have a follow-up coronary angiography performed according to current recommendations. However, the clinical analysis is not a major gaol of this study.

The investigators plan to evaluate following parameters:

* Whole blood morphology, creatinine, glucose, sodium, potassium, urea, lipid profile, CK, AST, fibrinogen, using standard methods in hospital laboratory.
* Inflammation markers - fibrinogen (nephelometry, Dade Behring) high-sensitivity C-reactive protein (nephelometry, Dade Behring); interleukin 6 (ELISA, R&D Systems).
* Thrombin generation markers in peripheral blood - thrombin-antithrombin complexes [TAT] (ELISA, Dade Behring); prothrombin fragments 1+2 [F1+2] (ELISA, Dade Behring).
* Fibrin clot permeation and susceptibility to lysis - measurement of Darcy's constant (dimensions of pores in the structure of the clot) by measurement of volume of buffer (0,05 mol/l Tris HCl with 0,15 mol/l NaCl) penetrating through the fibrin gel made in polystyrene pipes, 1.3 mm in diameter, with 100 ul of citrate plasma and after addition of 1U/ml human thrombin and 20 mmol/l calcium chloride in room temperature within 120 minutes according to methodology described by Mills and al.
* Fibrin gel turbidimetry - plasma mixed with Tris buffer prepared as mentioned above in 2:3 ratio, after addition 1 U/ml thrombin and 16 mmol/l calcium chloride will be analyzed in the UV spectrometer (wave length 405 nm). Following variables will be measured: initiation time, absorption increasing time and absorption value in plateau, approximately 10 minutes after addition of thrombin to the mixture. After 2 hours, spectrophotometry assessment of the clot will be performed (400 to 800 nm) to measure the pore size and thickness of fibrin fibers using the Carr equation modified by Wolberg. Then fibrinolysis of fibrin gel will be measured by means of turbidimetry. Another lysis assay based on the measurement of D-dimer levels in the effluent flowing through fibrin gels will be performed according to the method of Collet et al.
* Activation of the coagulation system in a "minimally modified blood" model according to Rand et al. Non-anticoagulated blood will be divided into 10 1-ml samples added to the tubes with TF and phospholipids, and then clotting will be stopped by an anticoagulant cocktail. In the supernatant samples, Western blotting and HPLC analysis of fibrinopeptides will be performed as described previously.

In 40 patients allocated at a random we will assess activation of coagulation system using the vascular injury model according to a procedure developed by us.

We will measure:

* Activation of prothrombin
* Conversion of fibrinogen to fibrin
* Activation of factor V and inactivation of factor Va
* Activation of factor XIII
* Activation of TAFI
* Thrombin generation

Genetic analysis The investigators will determine the PlA1 PlA2 polymorphism in the integrin β3 gene using the PCR technique in DNA samples collected from peripheral blood leukocytes.

Additionally, we are going to search for polymorphism of promoter region of IL-6 /G-174C also by means of PCR in DNA collected from peripheral blood leukocytes, using prim-ers 5'- AAT CTT TGT TGG AGG GTG AG and 5'- ACA TGC CAA GTG CTG AGT CA and restriction endonuclease Sfa NI on 2% agarose gel.

ELIGIBILITY:
Inclusion Criteria:

* Age < 75 years
* Acute coronary syndrome (symptom onset < 12 h)

Exclusion Criteria:

* Diabetes on insulin
* Anticoagulant therapy
* Renal insufficiency
* Liver injury
* Acute cardiovascular event within the previous 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
decrease in thrombin generation | 2 months

SECONDARY OUTCOMES:
increase in clot permeability | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Anetta Undas, Professor, Principal Investigator — Institute of Cardiology Jagiellonian University Krakow; Krzysztof Zmudka, Professor, Study Director — Insitute of Cardiology Jagiellonian University Krakow
Locations (1):
- Institute of Cardiology, Krakow, Poland

REFERENCES:
- [Derived] Undas A, Machnik A, Potaczek DP, Wypasek E, Zmudka K, Tracz W. Ezetimibe combined with simvastatin compared with simvastatin alone results in a greater suppression of oxidative stress and enhanced fibrinolysis in patients after acute coronary events. J Cardiovasc Pharmacol. 2011 Aug;58(2):167-72. doi: 10.1097/FJC.0b013e31821e8cb2. PMID 21558878